CLINICAL TRIAL: NCT05834608
Title: Cerebral Regional Oxygenation with Manual Versus Mechanical Ventilator Assisted Ventilation During Intravenous Induction in Pediatric Patients
Brief Title: Cerebral Regional Oxygenation with Manual Versus AutoFlow Ventilation
Status: Completed | Type: Observational
Sponsor: Marmara University (Other)
Responsible Party: Principal Investigator, Ruslan Abdullayev, Assoc. Prof., Marmara University
Other Study IDs: 09.2022.277
Record Dates: First submitted 2023-04-04; First posted 2023-04-28 (Actual); Last update posted 2024-12-31 (Actual); Status verified 2023-10

CONDITIONS: Oxygen Deficiency
MeSH Terms: conditions — Hypoxia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Group M: Manual ventilation
- Group A: AutoFlow mechanical ventilation
  Interventions: Behavioral: Mechanical ventilator-assisted ventilation

INTERVENTIONS:
Behavioral: Mechanical ventilator-assisted ventilation — After the intravenous anesthesia induction, mechanical ventilator-assisted ventilation with AutoFlow mode of the anesthesia machine (Draeger-Perseus) will be applied before intubation.
  Groups: Group A

SUMMARY:
Anesthesia induction is associated with hemodynamic imbalances that can affect the blood flow to major organs. Moreover it can result in deoxygenation as well. During standard anesthesia induction the patient is manually ventilated with a circle-valve-mask system until the effect of muscle relaxant shows of. Near-infrared spectroscopy (NIRS) is a modification of a well-known peripheral pulse oxymetry that is used in the detection of the regional oxygen saturation (rSO2) in organs, including brain, liver, muscle, and intestines. In this study we will compare the regional oxygenation status of the patients during anesthesia induction in which either standard manual ventilation or mechanical ventilator-assisted ventilation was performed. AutoFlow(R) mode of Draeger-Perseus mechanical ventilator will be used for the ventilator-assisted ventilation.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anaesthesiologists (ASA) physical status I-II

Exclusion Criteria:

* ASA III or above
* Congenital or traumatic brain injury
* Allergy to NIRS probe material
* Cardiac or vascular disease, including heart failure or hypertension
* Difficult mask ventilation and difficult intubation
* Thoracic surgery
* Head and neck surgery
* Emergency surgery
* Obesity

Ages: 5 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Pediatric surgical patients aged 5-10 years scheduled for elective surgery.
Sampling Method: Probability Sample
Enrollment: 51 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2023-01-01 (Actual); Study Completion 2023-08-04 (Actual)

PRIMARY OUTCOMES:
NIRS_-1 | 60 seconds before induction.
  Serebral oxygenation status measured by near-infrared spectroscopy device (INVOS oximeter, Somanetics, Troy, MI, USA).
NIRS_0 | At the start of anesthesia induction.
  Serebral oxygenation status measured by near-infrared spectroscopy device (INVOS oximeter, Somanetics, Troy, MI, USA).
NIRS_0.5 | 30 seconds after the anesthesia induction.
  Serebral oxygenation status measured by near-infrared spectroscopy device (INVOS oximeter, Somanetics, Troy, MI, USA).
NIRS_1 | 60 seconds after the anesthesia induction.
  Serebral oxygenation status measured by near-infrared spectroscopy device (INVOS oximeter, Somanetics, Troy, MI, USA).
NIRS_1.5 | 90 seconds after the anesthesia induction.
  Serebral oxygenation status measured by near-infrared spectroscopy device (INVOS oximeter, Somanetics, Troy, MI, USA).
NIRS_2 | 120 seconds after the anesthesia induction.
  Serebral oxygenation status measured by near-infrared spectroscopy device (INVOS oximeter, Somanetics, Troy, MI, USA).

CONTACTS AND LOCATIONS:
Overall Officials: Tumay Umuroglu, Prof. Dr., Principal Investigator — Marmara University Department of Anesthesiology and Reanimation
Locations (1):
- Marmara University School of Medicine, Istanbul, Pendik, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No